CLINICAL TRIAL: NCT05238701
Title: A Randomized, Double-blinded, Placebo-controlled, Dose-escalation Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetic of LPM3770164 Sustained-release Tablets in Healthy Subjects
Brief Title: A Dose-escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetic of LPM3770164 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03015/CT-CHN-101
Record Dates: First submitted 2022-01-09; First posted 2022-02-14 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Huntington Disease; Tardive Dyskinesia
MeSH Terms: conditions — Huntington Disease; Tardive Dyskinesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LPM3770164 (Experimental): LPM3770164 sustained-release tablets will be administrated with single dose from 0.5mg to 60mg
  Interventions: Drug: LPM3770164 sustained release tablet
- Placebo (Placebo Comparator): LPM3770164 sustained release tablet simulant will be administrated with single dose
  Interventions: Drug: LPM3770164 sustained release tablet simulant

INTERVENTIONS:
Drug: LPM3770164 sustained release tablet — LPM3770164 sustained release tablet will be administrated orally single-dose on day 1
  Other Names: LY03015
  Arms: LPM3770164
Drug: LPM3770164 sustained release tablet simulant — LPM3770164 sustained release tablet simulant will be administrated orally single-dose on day 1
  Other Names: LY03015 simulant
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blinded, placebo-controlled, dose escalation trial to evaluate the safety, tolerability and pharmacokinetic of LPM3770164 sustained-release tablets orally administered in healthy subjects under fasting state, providing the rationale information for subsequent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who voluntarily participate and sign the informed consent form;
2. Healthy male/female volunteers aged 18 to 45 years;
3. Body weight ≥ 50.0 kg for men and ≥ 45.0 kg for women, and body mass index (BMI) 18.5 ~ 28.0 kg/m2, inclusive;
4. Able to comply with the lifestyle restrictions.

Exclusion Criteria:

1. Subject has a history of allergy to any component of the investigational drug or similar drugs, or allergic constitution;
2. Subject has a current or past medical history that may affect the clinical trial or dysfunction, including but not limited to the past or current respiratory system, circulatory system, digestive system, urinary system, reproductive system, nervous system, endocrine system, immune system, motor system, blood system, psychiatry, dermatology and other clinically serious diseases or chronic diseases; or any other diseases that may interfere with the test results;
3. Any surgical condition or condition may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects;.
4. Subject has a history of self-mutilation; or at risk of suicide;
5. Subject has a history of surgery within 3 months prior to administration, or failure to recover from surgery, or having an expected surgical plan during the trial;
6. Subject has abnormal vital signs, laboratory abnormalities, and ECGs;
7. Subject has used any of over-the-counter products within 14 days or prescription medications within 28 days prior to dosing;
8. Subject positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab), or syphilis seroreactivity (Trust);
9. Subject has a history of alcohol abuse within 1 year or positive alcohol breath test results;
10. Subject has a history of substance abuse or a positive urine drug screen;
11. Subject who has daily smoking of ≥ 5 cigarettes;
12. Subject who has consumption of xanthine-rich foods or beverages (such as tea, coffee, cola, or chocolate) within 3 days prior to administration;
13. Subject who has consumption of food or beverages containing grapefruit within 7 days prior to administration;
14. Subject who has participated in other clinical trials within 3 months before administration;
15. Subject has used blood products or being blood donor or blood loss;
16. Pregnant, lactating women, or positive pregnancy test;
17. Subject who refusal to contraception, or plan to donate sperm or ovums;
18. Other conditions which would make participation in the study unsuitable.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2022-02-25 (Actual); Primary Completion 2023-11-04 (Actual); Study Completion 2023-11-04 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent adverse effects | from baseline to day 28
  Number of participants with treatment-emergent adverse effects will be summarized by Group, System Organ Classification (SOC), Preferred Term (PT), severity and the relationship with treatment.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) | from baseline to day 15
Time to maximum observed concentration (Tmax) | from baseline to day 15
Area under the concentration-time curve (AUC) | from baseline to day 15
Clearance (CL) | from baseline to day 15
Half-life (t1/2) | from baseline to day 15
Mean Residence Time (MRT) | from baseline to day 15
Haematology | baseline, day 3, day 8, day 15, day 28
Blood Chemistry | baseline, day 3, day 8, day 15, day 28
Urinalysis | baseline, day 15, day 28
Coagulation | baseline, day 15, day 28
Body Temperature | baseline, day 1, day 2, day 3, day 4, day 6, day 8, day 11, day 15, day 28
Respiratory Rate | baseline, day 1, day 2, day 3, day 4, day 6, day 8, day 11, day 15, day 28
Blood Pressure | baseline, day 1, day 2, day 3, day 4, day 6, day 8, day 11, day 15, day 28
Pulse Rate | baseline, day 1, day 2, day 3, day 4, day 6, day 8, day 11, day 15, day 28
Physical Examination | baseline, day 15, day 28
12 lead electrocardiogram corrected QT interval | baseline, day 1, day 2, day 3, day 4, day 6, day 8, day 11, day 15, day 28
Simpson-Angus Rating Scale (SAS) | baseline, day 3, day 28
Barnes Akathisia Rating Scale (BARS) | baseline, day 3, day 28
Abnormal Involuntary Movement Scale (AIMS) | baseline, day 3, day 28
Stanford Sleepiness Scale (SSS) | baseline, day 3, day 28

CONTACTS AND LOCATIONS:
Overall Officials: hufang Li, Doctor, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No